CLINICAL TRIAL: NCT00812266
Title: Randomized Phase III Trial of Topotecan and Cisplatin Versus Etoposide and Carboplatin in the Treatment of Patients With Previously Untreated Small Cell Lung Cancer and Extensive Disease
Brief Title: Topotecan and Cisplatin Versus Etoposide and Carboplatin in 1st Line Treatment of Patients With Small Cell Lung Cancer and Extensive Disease (SCLC-ED)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Danish Oncological Lung Cancer Group (Other)
Responsible Party: Principal Investigator, Seppo W. Langer, MD pHD, Danish Oncological Lung Cancer Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOLG7; DOLG7 (Other: Danish Oncological Lung Cancer Group Number)
Record Dates: First submitted 2008-12-19; First posted 2008-12-22 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Extensive Disease; First-Line; Small Cell Lung Cancer
Keywords: SCLC; Extensive disease; topotecan
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; Cisplatin; EC regimen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Topotecan + cisplatin
  Interventions: Drug: topotecan + cisplatin
- B (Active Comparator): Etoposide + carboplatin
  Interventions: Drug: Etoposide + carboplatin

INTERVENTIONS:
Drug: topotecan + cisplatin — topotecan IV 2 mg/sqm d1-3 + cisplatin IV 50 mg/sqm d3 q3W
  Arms: A
Drug: Etoposide + carboplatin — Etoposide 120 mg/sqm IV d 1-3 + carboplatin AUC 5 d1 q3W
  Arms: B

SUMMARY:
Randomised trial comparing standard chemotherapy with carboplatin and etoposide with a combination of topotecan and cisplatin in patients with inoperable lung cancer of small cell type.

DETAILED DESCRIPTION:
Fase III, multicenter randomised trial comparing up to six cycles of carboplatin and etoposide with up to six cycles of topotecan and cisplatin in patients with extensive stage small cell lung cancer and PS 0-3

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed SCLC
* Extensive stage
* No prior chemotherapy
* WHO PS 0-3
* Adequate organ function (liver, kidney)
* Adequate hematology (bone marrow)
* Informed consent

Exclusion Criteria:

* PS 4
* Inadequate organ function
* Uncontrolled infection
* Concomitant major medical contraindications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2006-01; Primary Completion 2013-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
2 years survival | 2 years

SECONDARY OUTCOMES:
Response rates | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Seppo W Langer, MD PhD, Principal Investigator — Dept. of Oncology, Rigshospitalet, Copenhagen
Locations (1):
- Dept. Oncology, Rigshospitalet, Copenhagen, Denmark